CLINICAL TRIAL: NCT06752421
Title: The Effect of Continuous Low Tidal Volume Ventilation During Cardiopulmonary Bypass on Postoperative Delirium: A Prospective Randomized Controlled Trial
Brief Title: Effect of Low Tidal Volume Ventilation on Postoperative Delirium
Acronym: CLEVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, MD, Associate Professor, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TABED-24-851
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Delirium (POD); Cardiopulmonary Bypass; Low Tidal Volume Ventilation; Cognitive Dysfunction, Postoperative
Keywords: Postoperative Delirium; Cardiopulmonary Bypass; low tidal volume ventilation; Cognitive Dysfunction
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: During cardiopulmonary bypass (CPB), apnea is routinely performed. In the control group, apnea ventilation will be continued, while in the intervention group, low tidal volume (LTV) ventilation will be applied.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Apnea (No Intervention): The apnea group serves as the control group. In routine Coronary Artery Bypass Grafting (CABG) surgery, after the cross clamp procedure, the mechanical ventilator is turned off, and the process is maintained by cardiopulmonary bypass (CPB). In this group, no mechanical ventilation will be provided after the cross clamp procedure, and apnea will be applied as part of routine care. The process will be entirely maintained by CPB.
- Group B: Low Tidal Volume (LTV) (Experimental): In the LTV group, mechanical ventilation will be maintained with low tidal volume parameters after the aortic cross-clamp procedure. This intervention includes a tidal volume of 3-4 mL/kg, respiratory rate of 12-14 breaths/min, PEEP of 5-8 cmH₂O, and FiO₂ of 50%. Minute ventilation (MV) will not exceed 12 L, and the parameters are adjusted according to ideal body weight. This group is designed to evaluate the protective effects of low tidal volume ventilation during surgery.
  Interventions: Procedure: Group B: Low tidal volume

INTERVENTIONS:
Procedure: Group B: Low tidal volume — In the LTV group, mechanical ventilation will be maintained with low tidal volume parameters after the aortic cross-clamp procedure. This intervention includes a tidal volume of 3-4 mL/kg, respiratory rate of 12-14 breaths/min, PEEP of 5-8 cmH₂O, and FiO₂ of 50%. Minute ventilation (MV) will not exceed 12 L, and the parameters are adjusted according to ideal body weight. This group is designed to evaluate the protective effects of low tidal volume ventilation during surgery.
  Arms: Group B: Low Tidal Volume (LTV)

SUMMARY:
This study aims to evaluate the effect of low tidal volume (LTV) ventilation during cardiopulmonary bypass (CPB) on postoperative delirium. It is hypothesized that the risk of delirium, which negatively impacts recovery following cardiac surgeries, can be reduced by improving cerebral perfusion and oxygenation through LTV. The study is designed as a prospective, randomized, controlled trial comparing delirium incidence, ICU stay duration, and 30-day mortality/morbidity rates between LTV and apnea groups. Primary outcomes will be assessed using the 3D-CAM method, while secondary outcomes include ICU stay duration and mortality/morbidity rates.

DETAILED DESCRIPTION:
Introduction and Objectives:

This protocol aims to evaluate the effect of low tidal volume (LTV) ventilation during cardiopulmonary bypass (CPB) on postoperative delirium. Postoperative delirium, commonly seen after cardiac surgeries, negatively impacts patient recovery. It is hypothesized that LTV reduces the risk of delirium by improving cerebral perfusion and oxygenation. The study objectives include comparing the incidence of delirium, ICU stay duration, and 30-day mortality/morbidity rates between groups.

Study Design and Methods:

This prospective, randomized, controlled trial will involve two groups: patients receiving LTV ventilation and those undergoing apnea during CPB. Inclusion criteria target CABG patients over 18 years of age, while exclusion criteria include emergent surgeries and cognitive impairments. Randomization will ensure balanced group allocation through computer-based methods. Mechanical ventilation parameters will follow standard protocols for both groups.

Measurements and Hypotheses:

The primary outcome is delirium, assessed using the 3D-CAM method, while secondary outcomes include ICU stay duration and 30-day composite mortality/morbidity rates. LTV ventilation is expected to reduce delirium incidence, shorten ICU stay, and lower mortality/morbidity rates. Statistical analyses will include multivariable models to account for potential confounding factors.

Substudies and Limitations:

The protocol includes two substudies to evaluate microcirculation and renal perfusion. Limitations may arise from the overlap of sedation effects with delirium symptoms, variations in surgical techniques, and potential data loss during patient follow-ups. Interim analyses are planned to assess the study's safety and effectiveness. The study will be conducted without external funding, adhering to routine clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* All male or female patients over the age of 18
* Patients undergoing planned cardiac surgeries including CABG
* Patients with an American Society of Anesthesiologists (ASA) physical status of II, III, or IV

Exclusion Criteria:

* Emergency surgeries will be excluded due to the high likelihood of non-compliance with the protocol and the potential lack of essential patient information.
* Surgeries requiring single-lung ventilation will be excluded as they may cause confusion in determining any effects of the intervention due to the inability to apply the study intervention and the differential treatment of the lungs.
* Patients who meet delirium criteria according to 3D-CAM measurements during the initial visit will be excluded.
* Patients with a life expectancy of less than 6 months or a history of psychiatric or neurological diseases (including depression, severe central nervous system depression, schizophrenia, epilepsy, Parkinson's disease, and Alzheimer's disease) will be excluded.
* Severe impairments such as blindness, severe deafness, or dementia that may hinder cognitive testing will be excluded.
* Patients using psychotropic or opioid medications, those with a history of delirium, or those with a history of alcohol abuse or withdrawal within the past 6 months will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium incidence | From the point where the RASS score evaluating wakefulness is -3, for a duration of 48 hours
  The main objective of the study is to compare the rates of postoperative delirium between patients who received low tidal volume (LTV) ventilation and those who were apnea-induced during CABG surgeries. This will be measured by the incidence of delirium, and it will be statistically analyzed to determine whether there is a significant difference between the two groups.

SECONDARY OUTCOMES:
Length of stay in the intensive care unit (ICU) | The duration will be recorded in hours, starting from the time of ICU admission to the time of discharge.
  The duration of postoperative ICU stay will be measured and compared between the groups.
30-day mortality rate | In the first 30 days after surgery
  Mortality (death from any cause) rate occurring within the first 30 days post-surgery will be compared between the two groups .
30-day morbidity rate | In the first 30 days after surgery
  morbidity (complications such as infections, cardiac events, respiratory failure, renal dysfunction, etc.) rate occurring within the first 30 days post-surgery will be compared between the two groups .

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No